CLINICAL TRIAL: NCT05934214
Title: Immune-related Adverse Events From Immune Checkpoint Inhibitor Characterization Using VigiBase, the WHO Pharmacovigilance Database: An Exploration of Adverse Event Patterns and Signal Detection.
Brief Title: EXploring Immune-related Adverse Events of Immune checkpoinT Inhibitors Using VigiBase, the WHO Pharmacovigilance Database
Acronym: EXIT
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut Curie (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, prof., Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-23-05
Record Dates: First submitted 2023-06-16; First posted 2023-07-06 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Immune-related Adverse Event; Immune Checkpoint Inhibitor-Related Myocarditis
Keywords: Immune checkpoint inhibitors
MeSH Terms: conditions — Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- immune-related adverse event reaction: Reports of identified immune-related adverse event reaction
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Reports associated with an an Immune checkpoint inhibitor with a status of "Suspect" or "Interacting"
  ICI will include the following list of FDA-apporved ICIs:
  nivolumab, pembrolizumab, cemiplimab, dostarlimab, durvalumab, atezolizumab, avelumab, ipilimumab, tremelimumab, relatlimab

SUMMARY:
This is an observational, retrospective pharmacovigilance study based on reports registered and transmitted in VigiBase®, the WHO's international database.

This study includes all reports identified as exposure to an ICI and suspect of inducing adverse drug reaction.

The aim of the study is to characterize immune-related adverse reactions associated with immune-checkpoint inhibitors, particularly their time-to-onset, co-occurence, factors associate with their over-report and fatality.

DETAILED DESCRIPTION:
Over the past ten years, immuno-oncology (IO) has gradually integrated the therapeutic arsenal of cancer treatment. CTLA-4, program-death 1 (PD1) and its ligand (PD-L1) and LAG3 were found to be major targets active in multiple tumor types. Immune checkpoint inhibitors (ICI) are antibodies blocking these targets and became a cornestone of cancer treatment.

This is an observational, retrospective pharmacovigilance study based on reports registered and transmitted in VigiBase®, the WHO's international database. VigiBase is managed by the Uppsala Monitoring Centre (UMC, Uppsala, Sweden) and contains about 30 million reports (as of Jan 2023) submitted by national pharmacovigilance centers since 1967.

The use of VigiBase® for pharmacovigilance analyses is not dependent on institutional review board approval. It is conditioned on institutional access provided and approved by the Uppsala Monitoring Centre. Since spontaneous reporting systems are based on anonymity and the process only requires patient non-opposition, no informed consent was requested to use VigiBase® in this study.

This study includes all reports associated with an ICI. The query is performed using the Medical Dictionary for Regulatory Activities (MedDRA), between January 1st 2008 (year of first report of ICI in VigiBase), and January 1st 2023. The analysis focused on reports suspected to be induced by an ICI (as opposed to concurrent use).

ELIGIBILITY:
Inclusion Criteria:

* Any report with an ICI "Suspect" or "Interacting" with the reported adverse drug reaction.

Exclusion Criteria:

* ICI not FDA approved
* No irAE identified in report

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any reports with an immune-related drug reaction attributed to an immune checkpoint inhibitor
Sampling Method: Probability Sample
Enrollment: 141630 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Factors associated with an increased rate of fatality among reports with an immune-related adverse event (irAE). | any report prior to january 2023
  Reports with a fatal outcome will be compared to reports with no fatal outcome. Odds ratio will be calculated to compare covariates potentially associated with an increase risk of fatality, including irAE type, cancer type reported, patient's age, gender, comorbidities, type of ICI or ICI combination and other treatments.

SECONDARY OUTCOMES:
Factors associated with an increased reporting of main irAE types | any report prior to january 2023
  Main irAEs are identified through MedDRA terms declared. For each irAE and each risk factors, an odds ratio will be calculated to assess a potential over-reporting. Factors evaluated will include but will not be limited to: cancer type, anticancer treatment type, socio-demographic variables (gender, age, country of reporting etc ...), year of reporting among others.
Time to onset for each irAE type | any report prior to january 2023
Rate of relapse with treatment rechallenge | any report prior to january 2023
  For each irAE, the rate (percentage) of irAE reccurence after treatment rechallenge.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris
  - CIC Paris-Est / Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: Undecided